CLINICAL TRIAL: NCT04555499
Title: A Validation Study of a Structured Diagnostic Examination of Patients With Suspected or Confirmed Stroke Resulting in a Stroke Score
Brief Title: A Diagnosis Study of a New Prehospital Strokeidentification Test, the PreHospitalt Ambulans Stroke Test (PreHAST), to be Used to Triage Patients With Suspected Stroke
Acronym: Pre-HAST
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Mia von Euler, Associate Professor, Karolinska Institutet
Other Study IDs: Pre-HAST
Record Dates: First submitted 2014-09-09; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: stroke pre hospital identification TIA; Patients with suspected stroke; Ability to give informed consent
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspected stroke: Patients with suspected stroke who are evaluated by paramedics
  Interventions: Other: Standardized neurological examination

INTERVENTIONS:
Other: Standardized neurological examination

SUMMARY:
The aim of the Pre-HAST study is to improve identification and triage of patients with suspected stroke in order to get the right patient to the right level of care as fast as possible. Furthermore, the scale is also intended to use follow stroke symptoms in emergency care. The test is more extensive then the FAST or Cincinatti Stroke Scale and is in some aspects similar to the NIHSS but is shorter, easier and faster to perform to improve interexaminator variability and improve validity in less trained personal. The test is intended for awake patients with suspected stroke

DETAILED DESCRIPTION:
PreHAST (PreHospital Ambulance Stroke Test)

* for suspected stroke in awake patients The following parameters are tested.

  1. Commands • Evaluates ability to understand verbal commands (impressive aphasia?) and to carry out complex commands (apraxia?)

     • Give the command: open and close your eyes! Grip your hand! (non-paretic side) 0 - two correct 2 - one or none correct
  2. Eye position • Evaluates involuntary deviation of the gaze (déviation conjugée?). If present, this implies a serious injury and thus 2 p are given.

     • Observ if the patient have the eyes trained to one direction unmotivated 0 - normal 2 - Patient gaze in one direction only or preferably
  3. Visual field

     * The test should be conducte in both left and right visual field simulatneously to evaluate both if hemianopsia and/or negelct are present. Both symptoms implieas a sever injury and thus 2 p are given
     * Look the patient in the eyes and wave in both visual fields simultaneously. Ask the patient to point at the hand or hands waving.

       0 - normal 2 - Only distinguishes one hand
  4. Facial palsy Ask the patient to smile 0 - normal 1 - one side of the mouth is hanging
  5. Arm paresis Is tested in lying or sitting position, one arm at the time. Start with the strongest arm. Lift the arm 45 degrees and ask the patient to keep in the position for 10 s. Count audible. If the patient can't lift the arm, assist.

     If the inability to keep the arm elevated is due to pain - score 0 Right Left 0 - can maintain the arm in postition for 10 s 1 - The arm drifts down from the initial position within 10 s but does not rely on support 2 - Falls down to support within 10 s or directly
  6. Leg paresis Test in lying or sitting position, one leg at the time. Start with the strongest leg. Lift the leg 30 degrees and ask the patient to keep in the position for 10 s. Count audible. If the patient can't lift the leg, assist.

     If the inability to keep the leg elevated is due to pain - score 0 Right Left 0 - can maintain the leg in position for 5 s 1 - The leg drifts down from the initial position within 5 s but does not rely on support 2 - Falls down to support within 5 s or directly
  7. Sensory (pain)

     * Evaluation of eventual loss of sensory function. It is important that pain is tested as not to miss a serious and not too uncommon type of stroke localized in the brain stem (Wallenberg´s syndrome).
     * Pinch the bend of the arms and legs, respectively. The stimuli shall be done simultaneously at the left and right side. Ask the patient if he/she can feel the stimuli in the same way on both sides. If the patient only registers stimuli on one side, 2 p are given.

       0 - normal

       1 - registers stimuli on both sides but less on one side 2 - Only registers the stimuli on one side
  8. Language • Evaluate if the patient has an understandable speech as stroke can cause both slurred speech (dysarthria) and affected ability to find words (aphasia). This test does not distinguish between dysarthria or dysphasia . Patient who does not speak at all (is mute) is given 2 p.

     * Ability to talk is noted during the examination. If uncertain, ask the patient to repeat: "the weather is pretty today" 0 - Normal 1 -Slight or moderate dysartria or aphasia. Communication possible. 2 - Severe dysarthria or aphasia. Communication basically not possible.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke

Exclusion Criteria:

* Unconscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected stroke using pre hospital services in region Skåne, Sweden or being admited to Södersjukhuset in Stockholm, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
stroke diagnosis | within 2 weeks of recrutiment
  The Pre-HAST is performed in the ambulance, in the emergency room or in the acute stroke ward. Final diagnosis of stroke and imaging data is matched to the findings in the Pre-HAST test

SECONDARY OUTCOMES:
neuroimaging findings of large vessel oclusion | within 3 months
  Imaging findings of examined patients are reviewed

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Pre hospital services in Skåne, Sweden, Hässleholm, Skåne County
  - Södersjukhuset, Stockholm

REFERENCES:
- [Result] Andsberg G, Esbjornsson M, Olofsson A, Lindgren A, Norrving B, von Euler M. PreHospital Ambulance Stroke Test - pilot study of a novel stroke test. Scand J Trauma Resusc Emerg Med. 2017 Apr 11;25(1):37. doi: 10.1186/s13049-017-0377-x. PMID 28399897